CLINICAL TRIAL: NCT05014178
Title: Kidney Sodium Functional Imaging: Evaluation of Kidney Medullary Sodium Content Using 23Na MRI in Kidney Disease
Brief Title: Kidney Sodium Functional Imaging
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Nephrologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 118638
Record Dates: First submitted 2021-08-14; First posted 2021-08-20 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Disease; Nephrolithiasis; ADPKD
Keywords: cortico-medullary gradient
MeSH Terms: conditions — Renal Insufficiency, Chronic; Nephrolithiasis; Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Complete blood count, urea, electrolytes, calcium, phosphate, 25-hydroxyVitamin D, CRP, glucose, intact PTH, creatinine, cystatin C, and osmolality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Adult CKD stage 1-5 participants: * Age greater than or equal to 18 years
  * Estimated GFR < 90 mL/min/1.73m²
  Interventions: Diagnostic Test: Sodium-23 MRI
- Adult transplanted participants: • Age greater than or equal to 18 years
  Interventions: Diagnostic Test: Sodium-23 MRI
- Adult dialysis participants: * Age greater than or equal to 18 years
  * More than 3 months duration of therapy
  Interventions: Diagnostic Test: Sodium-23 MRI
- Adult ADPKD: • Age greater than or equal to 18 years
  Interventions: Diagnostic Test: Sodium-23 MRI
- Adults treated for nephrolithiasis: • Age greater than or equal to 18 years
  Interventions: Diagnostic Test: Sodium-23 MRI
- Adult healthy controls including kidney donors: * Age greater than or equal to 18 years
  * Lack of kidney disease, heart failure, liver cirrhosis and peripheral
  Interventions: Diagnostic Test: Sodium-23 MRI

INTERVENTIONS:
Diagnostic Test: Sodium-23 MRI — Participants will lay in the MRI bed for approximately 60 minutes during scanning while the MRI technologist takes detailed pictures of their kidneys.

SUMMARY:
The corticomedullary gradient is largely responsible for developing the gradients that are needed to concentrate urine (more solutes and less water). The ability of the kidneys to produce concentrated urine is a major determinant of the ability to survive the warm weather. When temperatures are high, we lose water through sweat, and so the kidneys retain water to maintain fluidity in the blood. The maintenance of a sodium (salt) gradient is required for urine concentration because increased medullary sodium concentration increases the reabsorption of water into the kidney, to be redistributed in the blood. The purpose of this study is to know if the corticomedullary gradient is altered in patients across a wide spectrum of kidney disease using sodium Magnetic Resonance Imaging (MRI), a machine that takes pictures and measures the salt content in the kidneys. 23Na kidney MRI, will provide functional MR of the kidney as a non-invasive tool to describe medullary function to improve management of chronic and kidney disease.

DETAILED DESCRIPTION:
This study is a pilot exploratory study (preliminary project to assess the use of a kidney sodium coil across a wide spectrum of kidney disease). Approximately 200 patients from the London Health Sciences Regional Renal Program will be recruited. This study involves two visits at Robarts Research Institute or St. Joseph's Hospital, London, Ontario depending on scanner availability, lasting approximately 2 hours.

At the first study visit participants will undergo a sodium MRI scan of your kidneys. Prior to the scan, participants will have their sitting blood pressure and heart rate measured three times consecutively using a standard automatic blood pressure monitor. In addition to this, participants will be asked to provide a spot urine sample and have blood work done. If participants have been treated for nephrolithiasis, they will be responsible for completing a 24-hour urine volume test sometime the week before the MRI scan.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* For healthy controls: lack of kidney disease, heart failure, liver cirrhosis and peripheral edema
* For CKD stage 1-5: Estimated GFR < 90 mL/min/1.73m²
* For patients on maintenance hemodialysis or peritoneal dialysis: more than 3 months duration of therapy

Exclusion Criteria:

* Pregnant, breastfeeding or intending pregnancy
* Contraindication to MRI

  * Inability to tolerate MRI due to patient size and/or known history of claustrophobia.
  * Mechanically implanted, electrically, or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, tattoos, shunt, surgical staples (including clips or metallic sutures and/or ear implants.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CKD stage 1-5 Transplanted patients Maintenance dialysis (hemo and PD) ADPKD patient Patients treated for nephrolithiasis Healthy controls, including kidney donors
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Exploratory cortico-medullary gradient measurement | Throughout study visit, on average 2 hours
  Exploratory cortico-medullary gradient measurement in a large range of kidney disease by measuring sodium medullary to cortex ratio with23Na kidney MRI in:
  1) stage 1-5 CKD patients 2) transplanted patients 3) dialysis patients 4) ADPKD patients 5) nephrolithiasis patients (characteristically associated with salt loading) 6) healthy controls including kidney donors

SECONDARY OUTCOMES:
Urinary osmolarity | Throughout study visit, on average 2 hours
  To evaluate the relationship between sodium medullary to cortex ratio and urinary osmolarity
Renal Function | Throughout study visit, on average 2 hours
  To evaluate the relationship between sodium medullary to cortex ratio and renal function
Native and transplanted kidney | Throughout study visit, on average 2 hours
  To compare sodium medullary to cortex ratio between native kidney and transplanted kidney
Kidney biopsy | Throughout study visit, on average 2 hours
  To compare sodium medullary to cortex ratio between transplanted kidney and kidney biopsy
Residual renal function | Throughout study visit, on average 2 hours
  To evaluate sodium medullary to cortex ratio in dialysis patients and renal residual function
Nephrolithiasis | Throughout study visit, on average 2 hours
  To compare sodium medullary to cortex ratio between healthy control and patients who have nephrolithiasis
ADPKD | Throughout study visit, on average 2 hours
  To evaluate the ability to measure sodium medullary to cortex ratio in autosomal dominant polycystic kidney disease
Clinical practice | Throughout study visit, on average 2 hours
  To determinate if measurement of sodium medullary to cortex ratio measurement is meaningful in clinical practice

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Hospital, London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lemoine S, Akbari A, Brahm G, Dorie J, Tamasi T, Penny J, McIntyre CW. Redefining the concept of residual renal function with kidney sodium MRI: a pilot study. Nephrol Dial Transplant. 2024 Oct 30;39(11):1809-1816. doi: 10.1093/ndt/gfae070. PMID 38688870